CLINICAL TRIAL: NCT07003646
Title: Reperfusion Treatment in Acute Pulmonary Embolism: A Multicenter Observational Study in the Nordic Countries
Brief Title: Reperfusion Treatment in Acute Pulmonary Embolism
Acronym: PE-NORDIC
Status: Recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Stockholm South General Hospital (Other); Karolinska University Hospital (Other); Danderyd Hospital (Other); University Hospital, Linkoeping (Other); Sunderby Hospital (Other); Aarhus University Hospital (Other); Örebro University, Sweden (Other); Odense University Hospital (Other); Skane University Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kristina Svennerholm, Principal investigator. MD. PhD., Sahlgrenska University Hospital
Other Study IDs: PE-NORDIC
Record Dates: First submitted 2025-05-16; First posted 2025-06-04 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Embolism
Keywords: Thrombolysis; Catheter-directed intervention; Aspirational thrombectomy; Catheter-directed tromboylsis; High-risk PE
MeSH Terms: conditions — Pulmonary Embolism | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Catheter-directed intervention: Catheter-directed intervention, any device
  Interventions: Procedure: Catheter directed intervention, any device
- Systemic thrombolysis: Intravenous thrombolysis with tissue-type plasminogen activator (tPA)
  Interventions: Drug: Alteplase

INTERVENTIONS:
Procedure: Catheter directed intervention, any device — Catheter directed intervention for treatment of pulmonary embolism
  Groups: Catheter-directed intervention
Drug: Alteplase — Systemic thrombolysis
  Groups: Systemic thrombolysis

SUMMARY:
International guidelines recommend immediate reperfusion with systemic thrombolysis (ST) as first-line treatment in high-risk pulmonary embolism (PE). The therapy improves hemodynamics and overall survival but is also associated with a significant risk of severe bleeding. Catheter-directed intervention (CDI) is recommended as an alternative reperfusion therapy in high-risk PE when ST is contraindicated or has failed, as well as in patients who deteriorate or fail to improve during anticoagulation (AC) treatment. Despite lack of high-quality evidence and randomized studies between CDI and standard care, the use of CDI is spreading rapidly in high-risk PE and in less severe PE not fulfilling current treatment criteria.

DETAILED DESCRIPTION:
Several CDI methods are available, including mechanical thrombectomy (MT) and catheter-directed thrombolysis (CDT), but no method is currently recommended over the other. In Sweden, the MT device FlowTriever® (FT) was introduced in 2021 and has since then been the predominant method. Industry sponsored trials have investigated FT in uncontrolled observational trials and primarily in intermediate-risk PE. The investigator-initiated research on FT is limited to relatively small, descriptive, single-arm studies, or trials focusing on intermediate-risk PE.

There are several ongoing trials comparing different CDI methods to anticoagulation. However, in clinical practice, patients with acute PE may be subjected to different reperfusion strategies depending on severity and available resources. The PE-NORDIC observational study will compare the outcomes of different patient groups treated with current CDI methods used in the Nordic countries to patients treated with ST.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (≥18 years), including pregnant women, with verified (CTPA, angiography or scintigraphy) acute pulmonary embolism who are planned for, or have received, treatment with catheter directed intervention or systemic thrombolysis
* Informed consent (for patients who do not survive before informed consent can be obtained, a waiver of consent applies)

Exclusion Criteria:

* Ongoing enrolment in interventional catheter directed intervention trial
* Surgical embolectomy as primary reperfusion treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pulmonary embolism patients treated with catheter directed intervention or systemtic thrombolysis in hospitals in Sweden and Denmark where the former treatment modality is established.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Composite of severe bleeding or mortality at 30 days | From treatment to day 30 after treatment
  A composite of severe bleeding according to GUSTO (defined as intracranial bleeding or bleeding with substantial hemodynamic com-promise requiring treatment) or death within 30 days after treatment

SECONDARY OUTCOMES:
Mortality | 30 days
  Incidence of all-cause mortality
Mortality | 30 days
  Cause of death
Bleeding | 30 days
  Defined by GUSTO criteria, severe/non-severe.
Rescue treatment | 30 days
  Incidence of rescue treatment for PE (Systemic thrombolysis/Catheter-directed intervention/extracorporeal membrane oxygenation (ECMO)/surgical embolectomy)
Recurrent PE | 30 days
  Clinically relevant recurrence of PE
Hospital free days | 30 days
  Hospital free days between treatment and 30 days
ICU/HDU free days | 30 days
  Intensive care unit (ICU) and/or high dependency unit (HDU) free days between treatment and 30 days
Change in RV/LV ratio | 72 hours
  Change in right ventricular to left ventricular (RV/LV) diameter ratio before and within 72 h after treatment.
RV dysfunction | 1 year
  Examined by echocardiogram in association with follow-up visit 1 and 2
Persisting dyspnea | 1 year
  Self-reported level of dyspnea at follow-up visit 1 compared to discharge date and at follow-up visit 2 to compared to visit 1.
6-minute walk test | 1 year
  Distance (meters) walked in a 6-minute walk test performed at follow-up visit 1 and 2
Sit-to-stand 60 test | 1 year
  Number of stand-ups performed in a sit-to-stand 60 test performed at follow-up visit 1 and 2
PEmb-QoL | 1 year
  Pulmonary Embolism Quality of Life Questionnaire. Disease-specific health-related quality of life.
  FC: Frequency of complaints (8 items, reverse scoring where lower scores correspond to better quality of life).
  AD: Activities of daily living limitations (13 items, reverse scoring where lower scores correspond to better quality of life).
  WR: Work-related problems (4 items, reverse scoring where lower scores correspond to better quality of life).
  SL: Social limitations (1 item).
  IC: Intensity of complaints (2 items).
  EC: Emotional complaints (10 items, reverse scoring where lower scores correspond to better quality of life).
MRC dyspnoea scale | 1 year
  Medical research council dyspnoea scale. 0-4, a higher number corresponds to more dyspnoea.
EQ-5D-5L | 1 year
  EuroQol 5-dimension 5-level questionnaire. Generic health-related quality of life assessment.
  Movement (1-5), 1 corresponds to high and 5 to low movement level (descriptive)
  Care (1-5), 1 corresponds to high and 5 to low care level (descriptive)
  Activity (1-5), 1 corresponds to high and 5 to low activity level (descriptive)
  Pain (1-5), 1 corresponds to low and 5 to high pain level (descriptive)
  Anxiety (1-5), 1 corresponds to low and 5 to high anxiety level (descriptive)
  EQ-VAS (0-100), where 0 corresponds to worst health and 100 to best possible
PVFS scale | 1 year
  Post venous thromboembolism functional status scale (0-4) 0 corresponds to not affected of thromboembolism daily, 4 severely affected in daily life.
Incidence of CTEPH | 1 year
  Incidence of chronic thromboembolic pulmonary hypertension (CTEPH)
Cardiac biomarkers | 1 year
  Troponin and NTproBNP

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Svennerholm, Assoc Prof, Principal Investigator — Sahlgrenska University Hospital
Locations (13):
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- Sweden (10):
  - Sahlgrenska University Hospital, Gothenburg
  - Linköping University Hospital, Linköping
  - Sunderby Hospital, Luleå
  - Skåne University Hospital, Lund
  - Örebro University Hospital, Örebro
  - Danderyd Hospital, Stockholm
  - Karolinska University Hospital Huddinge, Stockholm
  - Karolinska University Hospital Solna, Stockholm
  - Södersjukhuset, Stockholm
  - Uppsala University Hospital, Uppsala

DOCUMENTS (2):
  • Study Protocol (2025-05-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT07003646/Prot_000.pdf
  • Statistical Analysis Plan (2025-07-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT07003646/SAP_001.pdf